CLINICAL TRIAL: NCT05527574
Title: Development of an Innovative Home-based Strategy for FrAilty preveNTion in AdultT With dIabetes and Chronic Kidney Disease (FANTASTIC)
Brief Title: Home-based Interventions for FrAilty preveNTion in AdultS With DIabeTes and Chronic Kidney Disease
Acronym: Fantastic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00089513
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Type 2; Frailty; Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Frailty; Kidney Diseases | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise Intervention Frail (Experimental): Resistance Exercise Intervention (home video education: resistance training and diet education) for Frail participants
  Interventions: Other: Resistance Exercise
- Standard of Care or Control Frail (No Intervention): Standard of Care (standard diet and physical activity education) for Frail Participants
- Exercise Intervention Pre-Frail (Experimental): Resistance Exercise Intervention (home video education: resistance training and diet education) for Pre-Frail participants
  Interventions: Other: Resistance Exercise
- Standard of Care or Control Pre-Frail (No Intervention): Standard of Care (standard diet and physical activity education) for Pre-Frail Participants

INTERVENTIONS:
Other: Resistance Exercise — Participants are enrolled in 30-40 minutes of resistance exercise training using elastic bands for 30-40 minutes/session three times per week over six months
  Arms: Exercise Intervention Frail; Exercise Intervention Pre-Frail

SUMMARY:
One of the most common problems in people with diabetes (DM) and chronic kidney disease (CKD) is the high frequency of other coinciding medical conditions such as osteoporosis and frailty. Frailty in particular is very common in adults with DM and CKD and it can result in significant muscle weakness which can result in increasing difficulties with performing activities of daily life (ADL). This can lead to an increase risk for falls, bone fractures and increasing hospitalization. The investigators have showed that adults with DM and CKD who have frailty use hospital services more frequently, have reduced quality of life and difficulties with performing their ADLs1. There is some evidence that early screening for frailty and lifestyle interventions that focus on healthier eating and physical activity can help prevent frailty from getting worse. The study purpose is to develop and test a home-based lifestyle intervention program focused on optimizing diet and the ability to perform your ADLs in adults with DM and CKD. The goal of this program is to ensure that adults with DM can live healthier lives within the community.

DETAILED DESCRIPTION:
Research Hypothesis: A home based video program focused on education related to lifestyle modification (diet, physical activity) over 6 months will result in improved measures of muscle strength/muscle functionality, health related quality of life and reduced measures of frailty and health care utilization in adults with DM and CKD.

V. Expected Outcomes: Results from this study will address two important questions a) identification of features of frailty/pre-frailty in adults with DM and CKD who should be targeted for lifestyle intervention b) development of home based programming for individuals with pre-frailty/frailty in the community dwelling adults with DM. This information is needed to help our clinical teams screen for frailty/pre-frailty and to focus health care resources on developing rehabilitation strategies to prevent and treat adults patients with DM and Frailty. This is particularly relevant for those who are 'vulnerable to Frailty' (pre-frail), but do not have the full condition. Prevention of the progression to full FRAILTY is critical to ensure optimal mental health HRQOL, to reduce health care use and to improve diabetes interventions in the community for those most vulnerable (Core Area 1). This will promote healthy aging in the community setting in obese adults with DM by supporting independent living, quality of life, mental health and delayed care utilization (Core Area 2) and will ensure healthy lives and promote well-being of all adults with DM at all ages (Goal 3).

Study Design:

There are two phases of this study. 1) Development of Video programming and 2) Open-label non-blinded study.

Phase 1 (see Table 1): Home Video content will be developed based on the principals of social cognitive theory. Video content will include two components a) resistance exercise (based on Canadian Diabetes Association video's that are adapted to meet the patient's functional capacity and b) the concepts of nutrition literacy. This will be done so a comprehensive approach to the lifestyle factors known to contribute to frailty (diet, exercise) can be developed in the educational programming of the video content (mp4 files). The resistance exercises will based upon Diabetes Canada resistance exercises which will have been adapted to meet the functional abilities of the patients in this population (based on the Investigator's earlier studies in DM and CKD) (Mager et al Can J Diabetes 2019) and https://www.diabetes.ca/getmedia/0a646e26-9e1c-4769-975f-51876edf6ecd/resistance-band-exercises-2.pdf.aspx ). Video content filming will be supported in the field by trained RA/graduate student and exercise specialists and then vetted for content and face validity by experts in the field (PT, MD, RD, geriatrician and exercise specialist CI and collaborators). We will also elicit patient feedback in vetting video content from participants from ongoing studies in the area (Pro00049292) and/or by recruiting potentially interested patients in the clinics. Participants who participate in this phase of the study will not be enrolled into Phase 2 of the study.

Table 1: Home Based Video Content (Mager/Manns/Boule/Juby) Phases Goals Nutrition Exercise Months:0-2

Training & Education Weight bearing and basic resistance exercise training

Optimizing Diet Quality (DQ) (glycemic control) Healthy Eating Carbohydrate counting Protein, Fat Micronutrients Weight bearing and balance activities: Establish routine walking activities. Goal setting/pace setting.

Resistance training: Elastic bands (1-2 sets/session) for 30 min x 3 times/wk Upper/lower limbs Months:2-4 Strength, Power & Endurance

DQ & Diet Diversity Increasing exercise endurance, power and training for weight bearing and resistance activities

Optimizing DQ (glycemic control, electrolyte status) Healthy Eating & Meal Preparation Sodium Potassium Phosphorus Glycemic Index Glycemic Load Weight bearing and balance activities (10 min sessions; 3 times weekly)

Resistance Activities:

Elastic bands (2-3 sets/session) for 30 minutes x 3 times weekly including upper/lower limbs Months 4-6 Maintenance

Nutrition Literacy Endurance, power activities for weight bearing, balance and resistance exercise.

Nutrition literacy/DQ Healthy Eating & Nutrition Literacy Food labels Grocery shopping Grocery Budgets Weight bearing/balance activities (10 minute session; 3-4 times weekly).

Resistance Activities: Elastic bands (3-4 sets/session) for 30 minutes x 3-4 times/week. Upper/lower limbs

Phase 2 Research Plan and Study Design: This is an open-label, non-blinded RCT. Participants will be recruited from the Diabetes Nephropathy Prevention Clinics (DNPC) and Renal Insufficient Clinics (RIC) in the Northern Alberta Renal Program (NARP) and undergo frailty screening by trained research personnel to determine frailty vs pre-frailty status using validated methodologies prior to randomization. Following this, the Investigators will randomize 120 participants (60/gp in blocks of frail vs non-frail) to one of two arms of the study: home based video intervention (n=60) or standard therapy (n=60) (diet/physical activity counseling) in a block design (frail (n=30/gp) vs pre-frail (n=30/gp)) at baseline (Figure 1).

Screening for frailty will be performed prior to randomization using the validated Clinical Frailty Scale; a tool widely used by clinicians to screen for frailty risk in many clinical populations. This tool takes approximately 5 minutes to administer and can be readily administered by trained research personnel in clinic. Study analysis will compare outcomes based on frail vs pre-frail in each group allocation (Frail (n=30) vs Pre-Frail (n=30); for a total of 60/group or 120 participants). The investigators will use a randomizer software (randomizer.org) to randomize study participants.

Study Visits: Visits to the Diabetes and Physical Activity Laboratory (DPAL)/Clinical Research Unit (CRU) at the University of Alberta will be made at baseline and 6 months for education related to study video technology/content (Table 1) and to perform study measurements related to frailty assessments, body composition, muscle strength, weight-bearing activity, HRQOL, mental health, cognition and anthropometrics . The Investigators will book DEXA scans at baseline and 6 months follow up with Medical Imaging Consultants; run by certified radiologists. There are two sites: one located within walking distance of the Clinical Research Unit, University of Alberta and one site located at Terra Losa, 9566- 170 Street, Edmonton AB. Education will include instruction re: video content on the electronic devices provided, review questionnaire content at baseline with weekly telephone calls to both groups in the first month to address questions. Home visits will be made q monthly by trained RA/graduate student to assess adherence to the prescribed therapies and to address concepts related to diet, nutrition literacy, and ALDs (Figure 1 and Table 1).

Figure 1: Study Design with primary and secondary outcomes

Standard of Care: This focuses on diet education aimed at promoting glycemic control (carbohydrate counting), electrolyte balance and increasing physical activity using Diabetes Canada and AHS Nutrition Education materials. Education related to physical activity is aimed at decreasing sedentary hours/increasing activity as per current Diabetes Canada Guidelines and Health Canada guidelines19. Participants randomized to the standard of care group will receive an accelerometer and will have monthly home visits by the RA to ensure equivalency of care in terms of the number of interactions with health care providers. This is necessary to reduce the risk for bias in study outcomes related to exposure to health care providers. This education will be conducted by a registered dietitian (RD) who is part of the research team. Participants will be provided with electronic devices as per Intervention group (questionnaires as per the intervention will be provided which will have standard educational materials uploaded on the devices.

Home Based Rehabilitation Intervention: Participants will be provided with a video (mp4 files) that will be uploaded to compatible portable electronic devices (such as tablets or lap tops). Tablets or other electronic devices will not require internet connections as the mp4 files will be uploaded on the devices prior to study start. Participants will listen and participate in video instruction for 3 times weekly (30-40 min; resistance exercise/balance/walking activities) and once/week for 15-20 minutes for nutrition based content. All exercises on the mp4 files will be performed by trained exercise specialists.

Questionnaires will be linked directly to each of the mp4 files on the electronic devices used for the instruction, ensuring that participants can directly answer validated questionnaires related to nutrition literacy (Self-Perceived Nutrition Literacy Scale 20), ADL independence (Barthel Index 21 and Lawton and Brody Scale 22 ) and food intake directly. This will make it simple and easy for participants to fill out questionnaires directly on the electronic devices where they viewed the home rehabilitation mp4 files. These will be filled out in the last week prior to the final visit by the team and then reviewed at the time of the visit. All data will be de-identified and answers from these scales will be downloaded onto a password protected-encrypted portable drive by the RA at the time of the home visit and/or via the internet (where available in the households).

Resistance training (RT) exercise; performed 3 times weekly for 30 minutes (Table 2): RT will be performed during the 6 months; 3 times/week in non-consecutive days for approximately 30 minutes sessions according to established guidelines. An additional 5 minute segments at the beginning/end of RT for warm-up/warm down will be provided. Programming and education will have an emphasis on patient participation in the RT programming to promote increased adherence. The RT will include the use of elastic bands. Elastic resistance provides similar prime mover, antagonist, assistant movers and stabilizer muscle activation as other forms resistance exercise in recreational users and have been validated in adults with frailty and are relatively inexpensive and easy to use.23 24 The elastic bands will be provided to study participants and instruction by an exercise specialist provided at the baseline visit.

RT routine: A circuit order of RT will be used for all major muscle groups; (Table 2). The order of the exercises will be randomly presented on the different mp4 files uploaded on the electronic devices to avoid an 'order effect' between individuals. Apps/icons on the electronic devices will be sufficiently large to ensure visual acuity and will be labelled to inform participant selection for weekly RT exercise.

ELIGIBILITY:
Inclusion Criteria:

* Adults (50-85 years)
* Clinically Diagnosed with diabetes (Type 2) and stage 1-IV CKD (Glomerular Filtration - Rate (GFR) 10-89 ml/min/1.73m2).

Exclusion Criteria:

* Functional and cognitive impairments (MMSE scores<24)
* Severe, permanent vision loss.
* Recent history of bone fracture in the last 12 months
* History of skeletal muscular disorders which precludes the ability to perform resistance exercises (e.g., moderate to severe osteoarthritis that prevents walking, bending and/or sit to stand or wheelchair dependent)
* Pregnant women
* Dialysis (hemodialysis or peritoneal dialysis) as treatment of kidney disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-08-22 (Estimated)

PRIMARY OUTCOMES:
Changes in frailty status in response to the exercise intervention | Six months
  Changes in frailty status (Edmonton Frailty Scoring System) in response to the home-based rehabilitation protocol vs standard of care over six months. Values in the Edmonton Frailty Scale range from 0-18 ; where values 0-5 are non-frail, 6-7 apparently frail vulnerable, 8-9 mild frailty, 10-11 moderately frail and 12-18 severely frail.

SECONDARY OUTCOMES:
Changes in total skeletal muscle mass surface area in response to exercise intervention | Six months
  Changes in total skeletal muscle area (total surface area/height square) (as measured by Dual X-ray Absorptiometry or DXA)
Changes in health related quality of life (HRQOL) | Six months
  SF-36; Short Form Health Survey; values range from 0-100 and will be compared with Canadian norms. Individual sub-domain scores (physical function, vitality, bodily pain, social function, role emotional, role physical, general health, mental health) and physical/mental composite scores. Each individual domain score and composite score ranges from 0-100; with Canadian age-sex matched reference data indicating values >80 as within healthy reference ranges.
Changes in cognitive health | Six months
  Mini-Mental State Examination (values > 26 are normal). No units.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Mager, PhD MSc RD, Principal Investigator — University of Alberta
Locations (1):
- Diabetic Nephropathy Prevention Clinic - Alberta Kidney Care - North, Edmonton, Alberta, Canada